CLINICAL TRIAL: NCT00154193
Title: A 12-month Study to Investigate the Correlations Between Cyclosporine Microemulsion C2 Levels (High, Medium and Low) and AUC0-4 With Regard to Outcome in de Novo Heart and Lung Transplantation - Identification of Target Cyclosporine Microemulsion C2 Levels.
Brief Title: Nordic Study in Cardiac and Lung Transplantation: Outcome in Relation to Cyclosporine Microemulsion C2 Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COLO400ANO01
Record Dates: First submitted 2005-09-06; First posted 2005-09-12 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2016-04

CONDITIONS: Heart and Lung Transplant
Keywords: Heart transplant, lung transplant, renal function, cyclosporine C2 Levels
MeSH Terms: interventions — Cyclosporine

ARMS (1):
- Cyclosporine (Active Comparator)
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: cyclosporine — patients will receive maintenance triple immunosuppression according to local practice consisting of Sandimmun Neoral, MMF/ECMPA or azathioprin and steroids.

SUMMARY:
The main purpose of this study is to identify cyclosporine C2 levels during 12 months treatment , while cyclosporine microemulsion dosages are adjusted based on C0 cyclosporine blood samples, and retrospectively correlate C2 levels to outcome (renal function and incidence of acute rejections)

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a first heart or bilateral or single lung transplant
* Patients for whom a triple maintenance immunosuppressive therapy consisting of cyclosporine microemulsion, steroids and mycophenolate mofetil (MMF)/ enteric-coated mycophenolate sodium (EC-MPS ,(or azathioprine) is indicated.

Exclusion Criteria:

* Multi-organ transplants or previously transplanted organs
* Patients with the need of more than two cyclosporine microemulsion dosages per day

Other protocol-defined inclusion/exclusion criteria may applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2004-06; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The average number of treated acute cardiac and lung graft rejection per patient during the first 12 months post transplant
The measured Glomerular Filtration Rate (GFR) at 3 and 12 months post-transplant

SECONDARY OUTCOMES:
Incidence of treated acute rejections
Incidence of biopsy-proven acute cellular rejections
Patient and Graft survival rates

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Derived] Iversen M, Nilsson F, Sipponen J, Eiskjaer H, Mared L, Bergan S, Nystrom U, Fagertun HE, Solbu D, Simonsen S. Cyclosporine C2 levels have impact on incidence of rejection in de novo lung but not heart transplant recipients: the NOCTURNE study. J Heart Lung Transplant. 2009 Sep;28(9):919-26. doi: 10.1016/j.healun.2009.05.022. PMID 19716045